CLINICAL TRIAL: NCT06239883
Title: The Academic Research Project Studies the Relationship Between Obstructive Sleep Apnoea and the Occurrence of Nocturia.
Brief Title: This Research Project Studies the Relationship Between OSA and Nocturia.
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: 468/2021
Record Dates: First submitted 2024-01-12; First posted 2024-02-02 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Nocturia; Lower urinary tract symptoms; Voiding diary; Nocturnal polyuria
MeSH Terms: conditions — Sleep Apnea, Obstructive; Nocturia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with OSA: Patients with diagnosed OSA will be included in this study group.
  Interventions: Other: Voiding diary

INTERVENTIONS:
Other: Voiding diary — The patients with diagnosed OSA will be asked to fill in the voiding diary.

SUMMARY:
The main goal of the study is to explore the relationship between obstructive sleep apnoea and nocturia.

DETAILED DESCRIPTION:
The observation study will be performed on patients diagnosed with obstructive sleep apnoea. Patients will undergo routine examination for sleep apnoea and will be asked to fill in voiding diaries for 48 hours. The main goal of the study is to find whether there are any parameters of sleep apnoea associated with occurrence of the nocturia.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed obstructive sleep apnoea (OSA )
* Apnea-Hypopnea Index (AHI) > 15
* ability to fill in the voiding diaries
* signed informed consent

Exclusion Criteria:

* patients using diuretics
* patients with malignancies
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diagnosed moderate or severe obstructive sleep apnoea (AHI > 15).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in the parameters of sleep apnoea - (apnea-hypopnea index - AHI) | 3 months
  The change in parameters of sleep apnoea - apnea-hypopnea index (AHI) will be monitored from the baseline to the end of follow-up, before and after the treatment intervention for correction of obstructive sleep apnoea (OSA). The obtained data will be correlated with the information from the voiding diary.
  The apnea-hypopnea index (AHI) is the combined average number of apneas and hypopneas that occur per hour of sleep. According to the American Academy of Sleep Medicine (AASM) it is categorized into mild (5-15 events/hour), moderate (15-30 events/hour), and severe (> 30 events/hour).ollow-up, before and after the treatment intervention for correction of obstructive sleep apnoea (OSA). The obtained data will be correlated with the information from the voiding diary.
Change in the parameters of sleep apnoea - oxygen desaturation index (ODI) | 3 months
  The change in parameters of sleep apnoea - oxygen desaturation index (ODI) will be monitored from the baseline to the end of follow-up, before and after the treatment intervention for correction of obstructive sleep apnoea (OSA). The obtained data will be correlated with the information from the voiding diary.
  ODI refers to the average number of desaturation episodes occurring per hour, where desaturation episodes are defined as a decrease in the mean oxygen saturation of ≥3% (over the last 120 seconds) that lasts for at least 10 seconds.
Change in the parameters of sleep apnoea - time under 90% saturation (T90) | 3 months
  The change in parameters of sleep apnoea - time under 90% saturation (T90) will be monitored from the baseline to the end of follow-up, before and after the treatment intervention for correction of obstructive sleep apnoea (OSA). The obtained data will be correlated with the information from the voiding diary.
  T90 was defined as the proportion of cumulative sleep time with oxygen saturation below 90% in total sleep time. T90≤5% of the total sleep time was classified as light hypoxia, T90 of 5-10% as mild hypoxia,10-25% as moderate hypoxia, and >25% as severe hypoxia.

SECONDARY OUTCOMES:
Change in the data from the voiding diary - functional capacity of the bladder | 3 months
  The change in bladder-derived parameters will be monitored from the baseline to the end of follow-up - functional capacity of the bladder will be measured in milliliters (mL).
Change in the data from the voiding diary - daily diuresis | 3 months
  The change in bladder-derived parameters will be monitored from the baseline to the end of follow-up - daily diuresis will be measured in milliliters (mL).
Change in the data from the voiding diary - number of voiding episodes | 3 months
  The change in bladder-derived parameters will be monitored from the baseline to the end of follow-up - the number of voiding episodes during sleep will be counted and monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Radek Paus Sýkora, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data with other researchers.

REFERENCES:
- [Background] Berry RB, Brooks R, Gamaldo C, Harding SM, Lloyd RM, Quan SF, Troester MT, Vaughn BV. AASM Scoring Manual Updates for 2017 (Version 2.4). J Clin Sleep Med. 2017 May 15;13(5):665-666. doi: 10.5664/jcsm.6576. No abstract available. PMID 28416048
- [Background] Lowenstein L, Kenton K, Brubaker L, Pillar G, Undevia N, Mueller ER, FitzGerald MP. The relationship between obstructive sleep apnea, nocturia, and daytime overactive bladder syndrome in women. Am J Obstet Gynecol. 2008 May;198(5):598.e1-5. doi: 10.1016/j.ajog.2008.02.024. PMID 18455544
- [Background] Oztura I, Kaynak D, Kaynak HC. Nocturia in sleep-disordered breathing. Sleep Med. 2006 Jun;7(4):362-7. doi: 10.1016/j.sleep.2005.10.004. Epub 2006 Mar 24. PMID 16564213
- [Background] Umlauf MG, Chasens ER, Greevy RA, Arnold J, Burgio KL, Pillion DJ. Obstructive sleep apnea, nocturia and polyuria in older adults. Sleep. 2004 Feb 1;27(1):139-44. doi: 10.1093/sleep/27.1.139. PMID 14998251
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434